CLINICAL TRIAL: NCT02859740
Title: Validation of the SIGAM/VF Mobility Grade
Acronym: SIGAM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GREMEAUX JOUSSAIN 2013-3
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- permanent prosthesis
  Interventions: Other: SIGAM Questionnaire
- Temporary prosthesis
  Interventions: Other: SIGAM Questionnaire

INTERVENTIONS:
Other: SIGAM Questionnaire

SUMMARY:
The objective of this study is to demonstrate the validity, the reproducibility and the coherence of the French version of the Special Interest Group in Amputee medicine (SIGAM) mobility scale questionnaire in adults with lower-limb amputations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Patients who have been informed about the research
* Patients with national health insurance cover
* Patients who accepted to take part in the study
* Able to understand simple instructions
* With transtibial, femoral, or bilateral amputation of the lower limb
* Whatever the etiology
* Patients able to do the 2-minute walk test
* Group 1:

  * Patients in the stabilized phase of the definitive prosthesis, with no modification of the prosthesis in the previous 3 months and at more than 6 months after the amputation.
* Group 2:

  * Patients in the initial phase of management (temporary prosthesis, rehabilitation) post trans-tibial unilateral amputation

Exclusion Criteria:

* Patient without national health insurance cover.
* Patients under guardianship.
* Pregnant or breast-feeding women.
* Alteration of executive functions making understanding of and compliance with the research protocol impossible (Mini Mental State Examination<20)
* Associated chronic motor deficiency, of neurological origin (examples: sequelae of stroke, balance and coordination disorders), or of osteo-articular origin (examples: knee or hip osteoarthritis), or due to secondary functional repercussions making it impossible to walk with a prosthesis.
* Severe medical disorder that significantly impairs functional capacities (severe heart failure, respiratory failure, non-stabilized metabolic disorders such as progressive kidney failure) that is life-threatening in the short or medium term (Progressive neoplastic disease, non-stabilized systemic disease).
* Complications at the stump other than microcirculation that could affect the application of a contact socket/sleeve: haematoma, Cysts, effusion, calcifications of soft tissues, bone spurs, infection (skin, abscess), neuroma, deterioration of the knee of the amputated limb, specifically painful Farabeuf angle (compression between bone and skin), venous thrombosis, abnormal stump shape making it impossible to use a socket (flexion of the knee, "pear-shaped", "deep-scar" stump…)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with temporary or permanent prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Answers to the SIGAM mobility scale questionnaire | Change from baseline at Week 2 and Week 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France